CLINICAL TRIAL: NCT04103996
Title: Incidence, Risk Factors and Outcomes of Diaphragm Dysfunction After Lung Transplantation
Acronym: RADAR
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-5894
Record Dates: First submitted 2019-08-27; First posted 2019-09-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diaphragm Injury; Lung Transplant; Complications, Mechanical; Respiratory Failure; Mechanical Ventilation Complication
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Sonographic measurements (diaphragm, abdominal muscle, and quadriceps thickness) will be acquired when listed for lung transplantation. Sonographic measurements will be recorded on a daily basis for up to 1 week after transplantation (while the patient remains intubated).
Diagnostic Test: Respiratory function measurements — Maximal expiratory pressure (MEP) and maximal inspiratory pressure (MIP) will be acquired after listing for lung transplantation. After transplant, MIP will be recorded once patients are eligible for a trial of spontaneous breathing and weekly thereafter. MEP will also be recorded at ICU discharge.

SUMMARY:
The study is designed to characterize the changes in diaphragm function after lung transplantation.

DETAILED DESCRIPTION:
Diaphragm dysfunction (DD) is a well-known complication after lung transplantation. Patients with an injured and dysfunctional diaphragm have greater difficulty weaning from mechanical ventilation post-transplant - they become too weak to breathe. However, little is known about the pre-transplant predictive factors associated with diaphragm dysfunction . We have developed a new technique employing beside ultrasound to measure diaphragm thickness. This allows us to observe changes in diaphragm muscle structure and function.

The goal of the study is to determine whether pre-transplant diaphragm thickness and function are associated with diaphragmatic dysfunction after lung transplantation. This will help us to confirm the best way to avoid diaphragm injury and to understanding the meaning of diaphragm ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than 18 years of age
* Listed for lung transplantation

Exclusion Criteria:

* Known diagnosis of chronic neuromuscular disease
* Relisting for transplantation
* Bridging to lung transplantation with respiratory support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enroll a total of 100 patients who were listed and will benefit from lung transplant
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of diaphragm dysfunction at the first spontaneous breathing trial and at ICU discharge after lung transplantation | First spontaneous breathing trial, an average of 1 to 7 days
  Diaphragm ultrasound will be used to visualize diaphragm dysfunction (maximal thickening fraction <20%)

SECONDARY OUTCOMES:
Pre-transplant diaphragm thickness and function compared to post-transplant diaphragm dysfunction | 1 day
  Diaphragm thickness and function documented on ultrasound will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — UHN Toronto
Locations (1):
- Toronto General Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No